CLINICAL TRIAL: NCT03331263
Title: Single Dose Pharmacokinetic Study to Assess the Systemic Exposure of Chlorhexidine From ReadyPrep® CHG (2% Chlorhexidine Gluconate Cloth)
Brief Title: Single Dose CHG Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: R17-023
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2021-04

CONDITIONS: Surgical Skin Preparation
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: laboratory-blinded, 3-period, 3-sequence, crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Abdominal application of 2% CHG (Experimental)
  Interventions: Drug: Chlorhexidine Gluconate
- Groin application of 2% CHG (Experimental)
  Interventions: Drug: Chlorhexidine Gluconate
- Control treatment with no application (No Intervention)

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — 2% CHG
  Arms: Abdominal application of 2% CHG; Groin application of 2% CHG

SUMMARY:
A single 2% topical application of ReadyPrep® CHG was applied on either the abdomen (Treatment-1) or the groin (Treatment-2) whereas Treatment-3 consisted of a control treatment where the same procedure as Treatment-1 and -2 was performed, but without the topical application of ReadyPrep® CHG. The treatments were separated by a wash-out of 7 calendar days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were male or female, aged ≥ 18 and ≤ 60 years (inclusive). The main inclusion criteria were:

  * non- or ex-smokers
  * body mass index (BMI) ≥19.00 kg/m2 and ≤32.00 kg/m2 and a body weight ≥ 55 kg
  * negative pregnancy test for female subjects
  * healthy according to medical history, complete physical examination (including vital signs and skin examination) and laboratory tests (general biochemistry, hematology and urinalysis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2017-08-06 (Actual); Study Completion 2017-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Carlson, Pharm D., Principal Investigator — Algorithme Pharma USA LLC
Locations (1):
- Algorithme Pharma USA LLC, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects were enrolled to participate in a 3-period, 3-sequence crossover study design
Pre-assignment Details: Each of the 12 subjects were scheduled to receive one of each treatment and randomized to what period they would receive each.
Groups:
- Control Treatment With no Application: No treatment
Period: Period 1
Arm/Group | Abdominal Application of 2% CHG | Groin Application of 2% CHG | Control Treatment With no Application
Started | 4 | 4 | 4
Completed | 4 | 4 | 4
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Abdominal Application of 2% CHG | Groin Application of 2% CHG | Control Treatment With no Application
Started | 4 | 3 | 4
Completed | 4 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Abdominal Application of 2% CHG | Groin Application of 2% CHG | Control Treatment With no Application
Started | 4 | 3 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were a total number of 12 subjects that started but only 10 subjects completed. Abdomen CHG application was completed on 12 subjects, Groin CHG application was completed on 10 subjects and control treatment was completed on 11 subjects.
Groups:
- All Study Participants: All 12 study participants are included
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Customized [Mean (Standard Deviation); unit: years] — >= 18 to <= 60 years of age (inclusive)
  years | 27 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 26 (3.3)
Weight (kg) [Mean (Standard Deviation); unit: weight in "kg"] | 75.6 (14.8)
Height (cm) [Mean (Standard Deviation); unit: cm] | 169.8 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasma Levels of Chlorexidine Following Systemic Exposure After a Single Topical Application of CHG.
Description: A total of 12 blood samples were collected (one tube of 6 mL each) at various time points up before and after product application in each study period and analyzed for plasma levels of chlorhexidine. Blood samples were collected at 10, 2 and 0.5 hours prior to each treatment, and 1, 2, 3, 4, 5, 6, 8, and 12 hours following each treatment.
Time Frame: Up to 24 hours after product application
Population: There was no statistical analysis planned on the PK results of this study. Results were reported as is. Study was completed as a 3-period, 3-sequence crossover therefore not all arms were analyzed with same amount of participants due to drop out.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Application of 2% CHG | Groin Application of 2% CHG | Control Treatment With no Application
Number analyzed (Participants) | 12 | 10 | 11
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With of Treatment Emergent Adverse Events.
Description: Number of subjects with treatment related adverse events as assessed by System Organ Class (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: Up to 24 hours after product application, overall, up to 3 weeks
Population: Study was completed as a 3-period, 3-sequence crossover therefore not all arms were analyzed with same amount of participants due to drop out.
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Application of 2% CHG | Groin Application of 2% CHG | Control Treatment With no Application
Number analyzed (Participants) | 12 | 10 | 11
Participants | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Three weeks
Arm/Group | Abdominal Application of 2% CHG | Groin Application of 2% CHG | Control Treatment With no Application
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 1/10 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abdominal Application of 2% CHG (N=12) | Groin Application of 2% CHG (N=10) | Control Treatment With no Application (N=11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — Sore Throat
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — congestion
Application site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0) — itching at application site (right groin)
Application site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Burning at application site (right groin)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written consent must be obtained

DOCUMENTS (1):
  • Study Protocol (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT03331263/Prot_000.pdf